CLINICAL TRIAL: NCT02946515
Title: Virtual Role-Plays to Reduce the Occurrence of Childhood Obesity
Brief Title: The SIM-PLICITY Study: The SIMulation Project - LIstening & Intervention in Pediatric obeSITY
Acronym: SIM-PLICITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: SIMmersion, LLC (Industry); University of Minnesota (Other); Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R44DP005954 (NIH); R44DP005954 (NIH)
Record Dates: First submitted 2016-10-25; First posted 2016-10-27 (Estimated); Results first posted 2019-08-26 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2017-07

CONDITIONS: Childhood Obesity
Keywords: Pediatrics
MeSH Terms: conditions — Pediatric Obesity | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Intervention (Experimental): The educational intervention will be the online simulation training program. Participants will be taught how to use the simulation during a 30 minute orientation session with a research staff person. We will use a mastery based approach rather than prescribing an absolute number of hours participants need to play. The criteria are as follows: 1) achieving a score of 90% or more on 2 out of the last 3 simulations played or 2) maximum of 8 hours of play, whichever comes first. After the orientation sessions, training sessions will be completed by participants on their own. The research team will confirm remote usage, and contact participants by email and phone to prompt usage as needed. The research team anticipates that the proposed method will accommodate for participant schedules while still ensuring intervention compliance.
  Interventions: Behavioral: Educational Intervention
- Waitlist Control Group (Experimental): The control group will participate in pre- and post-test assessments of their conversational skills with a trained actor. At the end of the study, the waitlist control group will be allowed to access to the simulation and the study team will provide training to participants upon request.
  Interventions: Behavioral: Wait List Control

INTERVENTIONS:
Behavioral: Educational Intervention — The educational intervention will be the online simulation training program. Participants will be taught how to use the simulation during a 30 minute orientation session with a research staff person. We will use a mastery based approach rather than prescribing an absolute number of hours participants need to play. The criteria are as follows: 1) achieving a score of 90% or more on 2 out of the last 3 simulations played or 2) maximum of 8 hours of play, whichever comes first. After the orientation sessions, training sessions will be completed by participants on their own. The research team will confirm remote usage, and contact participants by email and phone to prompt usage as needed. The research team anticipates that the proposed method will accommodate for participant schedules while still ensuring intervention compliance.
  Arms: Educational Intervention
Behavioral: Wait List Control — Access to the online simulation training after the follow-up measurement visit is complete
  Arms: Waitlist Control Group

SUMMARY:
This study is looking at the feasibility and efficacy of using SIMmersion's PeopleSim technology to train providers through role playing simulations to effectively conduct discussions with parents to provide intervention for, and reduce the likelihood of progression to childhood obesity.

DETAILED DESCRIPTION:
The prevalence of childhood obesity has tripled within the last twenty-five years (Skelton et al., 2009). Interventions targeting children are a high priority because children bear the greatest lifetime health risk from overweight and obesity (Ogden et al., 2007; Franks et al., 2010). Health professionals in primary care settings have the potential to reach large numbers of parents and children and address obesity because they have regular interactions with and are influential in the lives of families. Studies show that even brief advice delivered well can have a meaningful impact. To support providers in this important role, the Centers for Disease Control and Prevention collaborated with other health organizations to develop recommendations for assessment, prevention, and treatment of childhood and adolescent overweight and obesity. Despite the 2007 publication of these recommendations and increasing recognition of childhood obesity as a public health problem, rates of provision of obesity-related guidance and counseling remain low (Tanda & Salsberry, 2013), and research indicates that health care providers could use additional education, training, and support related to obesity prevention and treatment. Thus, effective strategies to support pediatric primary care providers in their efforts to intervene against address childhood obesity are needed. Building off the successes achieved in their Phase I study, SIMmersion LLC, in collaboration with Dr. Nancy Sherwood from HealthPartners Institute , Dr. Jayne Fulkerson from the University of Minnesota, and Dr. Michael Fleming from Northwestern University, will expand the Phase I simulation prototype, utilizing feedback provided by a team of independent experts. The innovative computer-based training system with interactive role-play simulations will provide health care providers with much needed experiential opportunities to develop skills in conducting discussions with parents and children about obesity. The product's efficacy will be evaluated in a randomized controlled trial (RCT); 100 pediatric, family practice, and nursing clinicians and trainees at various levels of experience will be recruited to participate. Half of the participants will be randomly assigned to the intervention group during which they will use the newly developed simulation product to develop their skills and half of participants will be randomly assigned to the wait-list control group; the primary outcome is performance in a role play with trained actors at 2 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older
* A health care provider within the HealthPartners Medical Group system or Park Nicollet clinic system OR a resident in the University of Minnesota pediatrics and family medicine residency program OR a student in the University of Minnesota nursing program or medical school
* Willing and able to participate in measurement visits and intervention activities
* See pediatric patients greater than or equal to 1/3 of their practice time

Exclusion Criteria:

* < 21 years of age
* Unable to ensure commitment to study measurement and intervention activities
* See pediatric patients less than 1/3 of their practice time

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E Sherwood, Ph.D, Principal Investigator — University of Minnesota
Locations (1):
- HealthPartners Institute, Bloomington, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fleming M, Olsen D, Stathes H, Boteler L, Grossberg P, Pfeifer J, Schiro S, Banning J, Skochelak S. Virtual reality skills training for health care professionals in alcohol screening and brief intervention. J Am Board Fam Med. 2009 Jul-Aug;22(4):387-98. doi: 10.3122/jabfm.2009.04.080208. PMID 19587253
- [Background] Kubik MY, Story M, Davey C, Dudovitz B, Zuehlke EU. Providing obesity prevention counseling to children during a primary care clinic visit: results from a pilot study. J Am Diet Assoc. 2008 Nov;108(11):1902-6. doi: 10.1016/j.jada.2008.08.017. PMID 18954581
- [Background] Story MT, Neumark-Stzainer DR, Sherwood NE, Holt K, Sofka D, Trowbridge FL, Barlow SE. Management of child and adolescent obesity: attitudes, barriers, skills, and training needs among health care professionals. Pediatrics. 2002 Jul;110(1 Pt 2):210-4. PMID 12093997
- [Background] Resnicow K, Davis R, Rollnick S. Motivational interviewing for pediatric obesity: Conceptual issues and evidence review. J Am Diet Assoc. 2006 Dec;106(12):2024-33. doi: 10.1016/j.jada.2006.09.015. PMID 17126634
- See also: Institutional Organization Website — http://www.healthpartners.com/institute/index.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medical and nursing students were recruited from a local university, and pediatric primary care practitioners were recruited through a local health system. All participants were recruited by email and invited to participate. Interested participants were contacted by study team members about the study and an in-person baseline visit was scheduled.
Pre-assignment Details: At baseline, participants reviewed and signed the consent form in-person and were given a hard copy for their records. After the baseline measurement visit, participants were randomized to either the intervention group or the wait-list control group. Due to the visit occurring in person, all participants who were consented were randomized (N=44).
Groups:
- Educational Intervention: The educational intervention was an online simulation training program. Participants were taught how to use the simulation during a brief phone orientation session with a research staff person. A mastery based approach was used, rather than prescribing an absolute number of hours participants need to play. The criteria were as follows: 1) achieving a score of 90% or more on 2 out of the last 3 simulations played or 2) maximum of 8 hours of play, whichever comes first. After the orientation sessions, training sessions were completed by participants on their own. The research team confirmed remote usage and contacted participants by email and phone to prompt usage as needed.
  The intervention group participated in pre- and post-test assessments of their conversational skills with a trained actor.
- Waitlist Control Group: The control group participated in pre- and post-test assessments of their conversational skills with a trained actor. At the end of the study, the wait-list control group were allowed to access to the simulation. Access was provided by the study team to all participants in the control group after completion of their post-test assessment.
Period: Overall Study
Arm/Group | Educational Intervention | Waitlist Control Group
Started | 22 | 22
Completed | 20 | 21
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Educational Intervention | Waitlist Control Group | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 19 | 33
  Male | 8 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 22 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 15 | 16 | 31
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Simulation Total Role Play Score
Description: Change from baseline in simulation total role-play score with a trained actor to evaluate the simulation's efficacy. The role-play scale measured the clinical skills of the participants assessed using standardized patients (SPs), blind to study condition, who acted as parents of a child with overweight during a well-child visit. Immediately following each 15-minute interaction with a study participant, the SP completed a checklist that assessed whether the participant 1) completed the skill correctly, 2) completed the skill incorrectly; or 3) did not complete the skill. Participants received a score of 1 if they completed the skill correctly in both Case A and Case B. The minimum score on the scale is 0 and the maximum score is 60, with higher scores indicating a better outcome.
Time Frame: 3 months after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Educational Intervention | Waitlist Control Group
Number analyzed (Participants) | 22 | 22
score on a scale
  Baseline Mean | 25.73 (6.27) | 23.73 (6.71)
  Follow-up Mean | 33.29 (4.75) | 25.89 (4.67)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Educational Intervention | Waitlist Control Group
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT02946515/Prot_SAP_000.pdf